CLINICAL TRIAL: NCT00442429
Title: Morbidity and Mortality Among Dialysis Patients After Treatment for Depression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Portland VA Medical Center (U.S. Federal Agency)
Collaborators: Medical Research Foundation, Oregon (Other)
Other Study IDs: 00898
Record Dates: First submitted 2007-03-01; First posted 2007-03-02 (Estimated); Last update posted 2007-03-02 (Estimated); Status verified 2007-03

CONDITIONS: Depression; ESRD
Keywords: depression; dialysis; kidney failure, chronic
MeSH Terms: conditions — Depression; Kidney Failure, Chronic; Renal Insufficiency; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Morbidity and Mortality among Dialysis Patients after Treating Depression

Objectives

Our investigation has two objectives:

1. To assess whether treatment and recovery from depression decreases adverse clinical events in chronic hemodialysis patients. Significant morbidity is associated with depression in dialysis patients, but subsequent impact on outcome after treatment of depression has not been reported.
2. To examine the rates of recovery from depression over a 6-month and 12-month period among prevalent dialysis patients. Rates of recovery among dialysis patients with depression are unclear. The natural history of depression among dialysis patients may help long-term management.

Plan and Methods

This project is a longitudinal prospective cohort study comprised of dialysis patients from outpatient dialysis units in the Portland, Oregon metropolitan area. Patients must be aged 18 or older and have started dialysis at least 90 days prior to enrollment. Patients are excluded if they are delirious, demented, cannot speak English, or have a prior psychiatric diagnosis other than depression. Baseline data collection includes patient demographics, etiology of renal disease, nutritional status, past medical and psychiatric history and baseline health status. Social support and quality of life assessments are obtained from direct interview. All patients are assessed for depression by the Beck Depression Index, a depression scale particularly useful in those with chronic illness, and the Diagnostic Interview Scale, a gold standard for depression assessment.

Those that are depressed will undergo pharmacologic treatment with an SSRI, if they agree, and be reassessed at 2 and 6 months for improvement. Patients who do not respond are referred for psychiatric therapy. The primary outcome of our study is the combined rate of prespecified morbidity and mortality at 18 months between two groups: depressed subjects agreeing to treatment and depressed subjects not agreeing to treatment. Prespecified morbidities include rates of 1) cardiovascular and cerebrovascular events, 2) infections, 3) vascular access complications, and 4) death. These were selected based on prior studies suggesting that depression increases cardiovascular and cerebrovascular events, suppresses the immune system, and up-regulates coagulation factors and platelet aggregation. , , , , , ,

Chi-square tests and T-tests will be used to compare baseline variables among those who are and are not depressed. A multivariable Cox proportional hazards model will compare survival among groups, with adjustments for baseline variables. Calculations derived from the Neyman-Pearson equation determined a sample size of 120 subjects.

Findings to date

We have enrolled 134 subjects to date, including 47 from the PVAMC, and 87 from outside dialysis units. Twenty-percent of them have been depressed. (We need to enroll 120 depressed patients.) No further results have been obtained this year. No further characteristics have been analyzed to date. All adverse events have been reported, none were unexpected.

Significance

We hope to demonstrate a reduction in adverse clinical outcomes with treatment of depression. If so, we would advocate that depression is a modifiable risk factor that warrants therapy for well-being in dialysis patients.

DETAILED DESCRIPTION:
Morbidity and Mortality among Dialysis Patients after Treating Depression

Objectives

Our investigation has two objectives:

1. To assess whether treatment and recovery from depression decreases adverse clinical events in chronic hemodialysis patients. Significant morbidity is associated with depression in dialysis patients, but subsequent impact on outcome after treatment of depression has not been reported.
2. To examine the rates of recovery from depression over a 6-month and 12-month period among prevalent dialysis patients. Rates of recovery among dialysis patients with depression are unclear. The natural history of depression among dialysis patients may help long-term management.

Plan and Methods

This project is a longitudinal prospective cohort study comprised of dialysis patients from outpatient dialysis units in the Portland, Oregon metropolitan area. Patients must be aged 18 or older and have started dialysis at least 90 days prior to enrollment. Patients are excluded if they are delirious, demented, cannot speak English, or have a prior psychiatric diagnosis other than depression. Baseline data collection includes patient demographics, etiology of renal disease, nutritional status, past medical and psychiatric history and baseline health status. Social support and quality of life assessments are obtained from direct interview. All patients are assessed for depression by the Beck Depression Index, a depression scale particularly useful in those with chronic illness, and the Diagnostic Interview Scale, a gold standard for depression assessment.

Those that are depressed will undergo pharmacologic treatment with an SSRI, if they agree, and be reassessed at 2 and 6 months for improvement. Patients who do not respond are referred for psychiatric therapy. The primary outcome of our study is the combined rate of prespecified morbidity and mortality at 18 months between two groups: depressed subjects agreeing to treatment and depressed subjects not agreeing to treatment. Prespecified morbidities include rates of 1) cardiovascular and cerebrovascular events, 2) infections, 3) vascular access complications, and 4) death. These were selected based on prior studies suggesting that depression increases cardiovascular and cerebrovascular events, suppresses the immune system, and up-regulates coagulation factors and platelet aggregation. , , , , , ,

Chi-square tests and T-tests will be used to compare baseline variables among those who are and are not depressed. A multivariable Cox proportional hazards model will compare survival among groups, with adjustments for baseline variables. Calculations derived from the Neyman-Pearson equation determined a sample size of 120 subjects.

Findings to date

We have enrolled 134 subjects to date, including 47 from the PVAMC, and 87 from outside dialysis units. Twenty-percent of them have been depressed. (We need to enroll 120 depressed patients.) No further results have been obtained this year. No further characteristics have been analyzed to date. All adverse events have been reported, none were unexpected.

Significance

We hope to demonstrate a reduction in adverse clinical outcomes with treatment of depression. If so, we would advocate that depression is a modifiable risk factor that warrants therapy for well-being in dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* ESRD age > 18

Exclusion Criteria:

* non english speaking, another psychiatric dx aside from depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 2004-07; Study Completion 2010-06

CONTACTS AND LOCATIONS:
Overall Officials: suzanne watnick, MD, Principal Investigator — PVAMC physician
Locations (1):
- Portland VA MC, Portland, Oregon, United States